CLINICAL TRIAL: NCT00440583
Title: Yt90 Zevalin & Combination Chemotherapy in Treating Patients With Stage II,Stage III,or Stage IV Diffuse Large B-cell Lymphoma
Brief Title: The Response Study of Yt90-Zevalin in Patients With Diffuse Large B-cell Lymphoma After 6 Cycles of CHOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH011101
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: CHOP-Z
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chemotherapy followed by Zevalin (Experimental): 6 cycles of chemotherapy with CHOP (Cyclophosphamide iv 750 mg/m2 over 15-45 minutes; Doxorubicin iv 50 mg/m2 over 5-20 minutes; and Vincristine iv 1.4 mg/m2 over 5-15 minutes on day 1 and oral prednisone 40 mg/m2 on days 1-5 repeated every 21 days), followed by Zevalin
  Interventions: Drug: chemotherapy followed by Zevalin

INTERVENTIONS:
Drug: chemotherapy followed by Zevalin — 6 cycles of chemotherapy with CHOP (Cyclophosphamide iv 750 mg/m2 over 15-45 minutes; Doxorubicin iv 50 mg/m2 over 5-20 minutes; and Vincristine iv 1.4 mg/m2 over 5-15 minutes on day 1 and oral prednisone 40 mg/m2 on days 1-5 repeated every 21 days), followed by Zevalin

SUMMARY:
The purpose of this study is to determine the effective of Yt90-Zevalin therapy in patients with diffuse large B-cell lymphoma that have achieved at least an unconfirmed partial remission after 6 cycles of CHOP therapy.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphomas (DLBCL) are the most common lymphoid neoplasm and account for 30% to 40% of adult non-Hodgkin lymphomas (NHL). DLCBL is a potentially curable disease. The ultimate goals of introducing new modality treatments such as monoclonal antibody (Ab)-targeted therapy are to increase complete remission (CR) rate and prolong event-free survival and overall survival.In phase II trials, it was shown that in DLBL the addition of rituximab to CHOP was feasible, with an increase in ORR, including CR and an increase in the OS and PFS in patients with DLBL.2 The benefit of R-CHOP was consistent across all subgroups of patients tested, including good and poor risks according to IPI and independent of younger than 70 years and older than 70 years of age.

Recently, new radiolabeled monoclonal antibodies have been established in the therapy of malignant lymphoma which can induce high remission rates. Radiolabeled antibodies are particularly effective as lymphoma cells are highly sensitive to radiation. In addition, the local emission of radiolabeled antibodies is able to destroy cells in close proximity to the bound antibody (bystander effect) therefore circumventing the problem of limited perfusion of bulky or poorly vascularized tumors.Ibritumomab is covalently linked to the tiuxetan chelate and radiolabeled with Yt90, producing Yt90-ibritumomab tiuxetan (Yt90-Zevalin). To optimize biodistribution, Rituximab is given prior to the radiolabeled antibody. Yt90-ibritumomab-tiuxetan-treatment was compared to a standard course of Rituximab. ORR in the Yt90-ibritumomab tiuxetan group was significantly higher than ORR in the Rituximab group (80% vs. 56% according to International Workshop Response criteria or 73% vs. 47% according to protocol-defined evaluation of response).

Since radioimmunotherapy represents a significant advance over unlabeled immunotherapy for the treatment of patients with B-cell non-Hodgkin's lymphoma, it is worthwhile to study the consolidation therapy with Yt90-ibritumomab tiuxetan (Yt90-Zevalin) in patients who achieved at least unconfirmed partial remission after 6 cycles of CHOP therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, CD 20 positive diffuse large B-cell lymphoma, meeting 1 of the following stage criteria: Bulky stage II disease, Stage III disease, Stage IV disease at the initial diagnosis.
* Bidimensionally measurable disease
* Age 18 - 75 Years
* Performance status Zubrod 0-2
* Less than 20,000/mcL circulating lymphoid cells on WBC differential count
* Adequate sections AND a paraffin block OR ≥ 10 unstained sections from the original diagnostic specimen available
* Needle aspiration or cytology are not considered adequate
* No clinical evidence of CNS involvement by lymphoma
* No prior diagnosis of indolent lymphoma
* No histologic transformation
* Life expectancy : Not specified
* Hepatic : Not specified
* Renal : Not specified
* Cardiovascular

  * Ejection fraction ≥ 45% by MUGA OR
  * No significant abnormalities by echocardiogram
* Pulmonary : No requirement for continuous supplemental oxygen
* Other

  * All adult patients of reproductive potential must use contraception during and for 6 months after completion of study treatment
  * No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, stage I or II cancer in complete remission, or carcinoma in situ of the cervix
  * No known HIV positive
* Written informed consent
* PRIOR CONCURRENT THERAPY:

  * Biologic therapy : No prior antibody therapy for lymphoma
  * Chemotherapy : 6 cycles of CHOP
  * Endocrine therapy : Not specified
  * Radiotherapy : No prior radiotherapy for lymphoma
  * Surgery : No prior solid organ transplantation

Exclusion Criteria:

* Previous antineoplastic treatment other than the 6 cycles of CHOP for the initial treatment of DLBCL
* Positive HIV serology
* Positive serology of HCV with the presence of HCV RNA of chronic hepatitis
* Positive serology of HBV with the presence of HBV RNA of chronic hepatitis
* Serum creatinine or bilirubin > 2.5 x upper limit of normal
* Active uncontrolled infection
* Concurrent severe and/or uncontrolled medical disease which could compromise the participation in the study
* Patients in whom more than 25% of the bone marrow has been infiltrated by lymphoma cells
* Patients with platelet counts <100,000/µl or neutrophil counts < 1500/µl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-09; Primary Completion 2011-09 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
- Determine the 2-years progression-free survival of consolidation therapy with Yt90-Zevalin. | 2 year

SECONDARY OUTCOMES:
Determine the response duration(time to progression)after therapy. | 2 year
Determine safety and tolerability of Yt90-Zevalin consolidation therapy. | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Surapol Issaragrisil, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand